CLINICAL TRIAL: NCT06202209
Title: The Impact of Autonomic Function on Recurrence Following Circumferential Pulmonary Vein Ablation for Atrial Fibrillation
Brief Title: The Impact of Autonomic Function on Atrial Fibrillation Recurrence After Pulmonary Vein Ablation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: China National Center for Cardiovascular Diseases (Other Government)
Collaborators: Xinjiang Uygur Autonomous Region Hospital of Traditional Chinese Medicine (Unknown); Xinjiang Corps Hospital (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2022-RW320-11
Record Dates: First submitted 2024-01-02; First posted 2024-01-11 (Actual); Last update posted 2024-01-11 (Actual); Status verified 2023-11

CONDITIONS: Atrial Fibrillation Recurrent
Keywords: Atrial Fibrillation Recurrent; Early recurrent atrial arrhythmia; Cardioneuroablation; Automatic function

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Circumferential Pulmonary Vein Isolation — Circumferential pulmonary vein isolation (CPVI) is a type of cardiac ablation procedure. Cardiac ablation procedures involve creating small scars in the heart using thermal or cold energy to block irregular electrical signals and restore normal heart rhythm. CPVI specifically creates small scars in the area where the four pulmonary veins connect to the left atrium of the heart. The pulmonary veins carry oxygen-rich blood from the lungs to the heart.

SUMMARY:
This is a prospective and observational study. The investigator speculated that the use of DC in patients with paroxysmal AF can serve as a predictor for early and late AF recurrence following CPVI.

DETAILED DESCRIPTION:
Atrial fibrillation (AF), also known as atrial flutter, is one of the most common cardiac arrhythmias and poses a serious threat to patients' health and well-being. The mechanism of AF is complex, with the autonomic nervous system playing a crucial role in its initiation and maintenance. Currently, medication and ablation are the main treatment methods to reduce AF episodes, but the efficacy of drug therapy is limited, and recurrence after ablation still exists. Recent studies have found that changes in autonomic nervous system activity are one of the key factors contributing to AF recurrence after ablation. Therefore, by objectively assessing changes in autonomic nervous system activity, it is expected to improve the success rate of AF ablation and provide a potential cure for AF, with significant social and economic value.

Studies have found that pulmonary vein isolation (PVI) ablation is the mainstream method for AF ablation, and it affects the autonomic nervous system function. Patients who show significant changes in autonomic nervous system function after AF ablation have higher success rates. Additionally, early-onset atrial arrhythmias are closely related to long-term AF recurrence after ablation. However, the mechanisms underlying early recurrence still require further investigation.

Our research team has conducted in-depth studies on the regulation of autonomic nervous system function in the heart and non-invasive assessment techniques, achieving breakthrough progress. The left atrial ganglion plays a crucial role in the initiation and maintenance of AF, and ablating the ganglion can improve the success rate of AF ablation. Non-invasive assessment techniques such as heart rate deceleration can quantitatively evaluate changes in vagal nerve activity in the heart, which can be used to predict the efficacy of autonomic ganglion intervention therapy.

Based on the above research, our research team hypothesizes that precise and quantitative assessment of autonomic nervous system function using heart rate deceleration can predict AF recurrence after PVI ablation. To validate this hypothesis, we plan to conduct a prospective observational study, recruiting patients with paroxysmal AF, assessing changes in autonomic nervous system function, monitoring early-onset atrial arrhythmias and AF recurrence, and providing theoretical support for the screening and intervention of high-risk recurrence patients, laying a foundation for clinical application.

ELIGIBILITY:
Inclusion Criteria:

1. Sign the informed consent form;
2. Clearly diagnosed as paroxysmal AF, willing to receive CPVI treatment;
3. A class I or class III antiarrhythmic drug with poor efficacy, or intolerance to drugs.

Exclusion Criteria:

1. Diagnosis of sinus rhythm at recruitment;
2. Age is <18 years old or> 75 years old;
3. Transthoracic echocardiography suggested a left atrial anterior and posterior diameter of> 55mm;
4. Previous history of catheter ablation or surgical ablation for AF;
5. Left atrial thrombus recorded by ultrasound or CT;
6. With severe pulmonary diseases;
7. Previous history of cardiac surgery;
8. Patients with hyperthyroidism, atrial septal defect, mitral valve stenosis or severe coronary heart disease who need further treatment;
9. During pregnancy or lactation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing CPVI due to paroxysmal atrial fibrillation.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-09-13 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-10-30 (Estimated)

PRIMARY OUTCOMES:
Recurrence of AF at 1 year after surgery | 12 months after CPVI
  Standard 12-lead surface electrocardiogram (ECG) and 24-hour ECG monitoring
Autonomic nerve function assessment | 12 months after CPVI
  The difference in DC values at 1 year compared to the preoperative baseline

SECONDARY OUTCOMES:
Recurrence of AF at 1 month after surgery | 1 months after CPVI
  Standard 12-lead surface electrocardiogram (ECG) and 24-hour ECG monitoring
Autonomic nerve function assessment | 1 months after CPVI
  The difference in DC values at 1 month compared to the preoperative baseline
Recurrence of AF at 3 months after surgery | 3 months after CPVI
  Standard 12-lead surface electrocardiogram (ECG) and 24-hour ECG monitoring
Autonomic nerve function assessment | 3 months after CPVI
  The difference in DC values at 3 months compared to the preoperative baseline

CONTACTS AND LOCATIONS:
Overall Officials: yan Yao, PhD, Study Chair — Fuwai Hospital,National Center for Cardiovascular Diseases
Locations (1):
- Fuwai Hospital, National Center for Cardiovascular Diseases, Chinese Academy of Medical Sciences and Peking Union Medical College, Beijing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Hindricks G, Potpara T, Dagres N, Arbelo E, Bax JJ, Blomstrom-Lundqvist C, Boriani G, Castella M, Dan GA, Dilaveris PE, Fauchier L, Filippatos G, Kalman JM, La Meir M, Lane DA, Lebeau JP, Lettino M, Lip GYH, Pinto FJ, Thomas GN, Valgimigli M, Van Gelder IC, Van Putte BP, Watkins CL; ESC Scientific Document Group. 2020 ESC Guidelines for the diagnosis and management of atrial fibrillation developed in collaboration with the European Association for Cardio-Thoracic Surgery (EACTS): The Task Force for the diagnosis and management of atrial fibrillation of the European Society of Cardiology (ESC) Developed with the special contribution of the European Heart Rhythm Association (EHRA) of the ESC. Eur Heart J. 2021 Feb 1;42(5):373-498. doi: 10.1093/eurheartj/ehaa612. No abstract available. PMID 32860505
- [Result] Staerk L, Sherer JA, Ko D, Benjamin EJ, Helm RH. Atrial Fibrillation: Epidemiology, Pathophysiology, and Clinical Outcomes. Circ Res. 2017 Apr 28;120(9):1501-1517. doi: 10.1161/CIRCRESAHA.117.309732. PMID 28450367
- [Result] Chen Z, Yang Y, Zou C, Zhang Y, Huang X, Li X, Yang X. Low heart deceleration capacity imply higher atrial fibrillation-free rate after ablation. Sci Rep. 2018 Apr 3;8(1):5537. doi: 10.1038/s41598-018-23970-7. PMID 29615802
- [Result] Sordillo LM, Redmond MJ, Campos M, Warren L, Babiuk LA. Cytokine activity in bovine mammary gland secretions during the periparturient period. Can J Vet Res. 1991 Jul;55(3):298-301. PMID 1716178
- [Result] Herring N, Kalla M, Paterson DJ. The autonomic nervous system and cardiac arrhythmias: current concepts and emerging therapies. Nat Rev Cardiol. 2019 Dec;16(12):707-726. doi: 10.1038/s41569-019-0221-2. Epub 2019 Jun 13. PMID 31197232
- [Result] Shen MJ, Choi EK, Tan AY, Lin SF, Fishbein MC, Chen LS, Chen PS. Neural mechanisms of atrial arrhythmias. Nat Rev Cardiol. 2011 Sep 27;9(1):30-9. doi: 10.1038/nrcardio.2011.139. PMID 21946776
- [Result] Shen MJ, Zipes DP. Role of the autonomic nervous system in modulating cardiac arrhythmias. Circ Res. 2014 Mar 14;114(6):1004-21. doi: 10.1161/CIRCRESAHA.113.302549. PMID 24625726
- [Result] January CT, Wann LS, Calkins H, Chen LY, Cigarroa JE, Cleveland JC Jr, Ellinor PT, Ezekowitz MD, Field ME, Furie KL, Heidenreich PA, Murray KT, Shea JB, Tracy CM, Yancy CW. 2019 AHA/ACC/HRS Focused Update of the 2014 AHA/ACC/HRS Guideline for the Management of Patients With Atrial Fibrillation: A Report of the American College of Cardiology/American Heart Association Task Force on Clinical Practice Guidelines and the Heart Rhythm Society. J Am Coll Cardiol. 2019 Jul 9;74(1):104-132. doi: 10.1016/j.jacc.2019.01.011. Epub 2019 Jan 28. No abstract available. PMID 30703431
- [Result] Ketels S, Houben R, Van Beeumen K, Tavernier R, Duytschaever M. Incidence, timing, and characteristics of acute changes in heart rate during ongoing circumferential pulmonary vein isolation. Europace. 2008 Dec;10(12):1406-14. doi: 10.1093/europace/eun287. Epub 2008 Oct 19. PMID 18936041
- [Result] Tang LYW, Hawkins NM, Ho K, Tam R, Deyell MW, Macle L, Verma A, Khairy P, Sheldon R, Andrade JG; CIRCA-DOSE Study Investigators. Autonomic Alterations After Pulmonary Vein Isolation in the CIRCA-DOSE (Cryoballoon vs Irrigated Radiofrequency Catheter Ablation) Study. J Am Heart Assoc. 2021 Feb;10(5):e018610. doi: 10.1161/JAHA.120.018610. Epub 2021 Feb 26. PMID 33634706
- [Result] Yang E, Ipek EG, Balouch M, Mints Y, Chrispin J, Marine JE, Berger RD, Ashikaga H, Rickard J, Calkins H, Nazarian S, Spragg DD. Factors impacting complication rates for catheter ablation of atrial fibrillation from 2003 to 2015. Europace. 2017 Feb 1;19(2):241-249. doi: 10.1093/europace/euw178. PMID 28172794
- [Result] Yao Y, Zheng L, Zhang S, He DS, Zhang K, Tang M, Chen K, Pu J, Wang F, Chen X. Stepwise linear approach to catheter ablation of atrial fibrillation. Heart Rhythm. 2007 Dec;4(12):1497-504. doi: 10.1016/j.hrthm.2007.07.028. Epub 2007 Aug 11. PMID 17997359
- [Result] Liang JJ, Elafros MA, Chik WW, Santangeli P, Zado ES, Frankel DS, Supple GE, Schaller RD, Lin D, Hutchinson MD, Riley MP, Callans DJ, Marchlinski FE, Dixit S. Early recurrence of atrial arrhythmias following pulmonary vein antral isolation: Timing and frequency of early recurrences predicts long-term ablation success. Heart Rhythm. 2015 Dec;12(12):2461-8. doi: 10.1016/j.hrthm.2015.07.015. Epub 2015 Jul 14. PMID 26187447
- [Result] Oral H, Knight BP, Ozaydin M, Tada H, Chugh A, Hassan S, Scharf C, Lai SW, Greenstein R, Pelosi F Jr, Strickberger SA, Morady F. Clinical significance of early recurrences of atrial fibrillation after pulmonary vein isolation. J Am Coll Cardiol. 2002 Jul 3;40(1):100-4. doi: 10.1016/s0735-1097(02)01939-3. PMID 12103262
- [Result] Nalliah CJ, Lim TW, Kizana E, Qian P, Kovoor P, Thiagalingam A, Ross DL, Thomas SP. Clinical significance of early atrial arrhythmia type and timing after single ring isolation of the pulmonary veins. Europace. 2015 Jul;17(7):1038-44. doi: 10.1093/europace/euu314. Epub 2015 May 2. PMID 25935165
- [Result] Zheng L, Yao Y, Zhang S, Chen W, Zhang K, Wang F, Chen X, He DS, Kadish AH. Organized left atrial tachyarrhythmia during stepwise linear ablation for atrial fibrillation. J Cardiovasc Electrophysiol. 2009 May;20(5):499-506. doi: 10.1111/j.1540-8167.2008.01371.x. Epub 2008 Nov 21. PMID 19054243
- [Result] Hu F, Zheng L, Liang E, Ding L, Wu L, Chen G, Fan X, Yao Y. Right anterior ganglionated plexus: The primary target of cardioneuroablation? Heart Rhythm. 2019 Oct;16(10):1545-1551. doi: 10.1016/j.hrthm.2019.07.018. Epub 2019 Jul 19. PMID 31330187
- [Result] Hu F, Zheng L, Liu S, Shen L, Liang E, Liu L, Wu L, Ding L, Yao Y. The impacts of the ganglionated plexus ablation sequence on the vagal response, heart rate, and blood pressure during cardioneuroablation. Auton Neurosci. 2021 Jul;233:102812. doi: 10.1016/j.autneu.2021.102812. Epub 2021 Apr 20. PMID 33940549
- [Result] Hu F, Zheng L, Liu S, Shen L, Liang E, Ding L, Wu L, Chen G, Fan X, Yao Y. Avoidance of Vagal Response During Circumferential Pulmonary Vein Isolation: Effect of Initiating Isolation From Right Anterior Ganglionated Plexi. Circ Arrhythm Electrophysiol. 2019 Dec;12(12):e007811. doi: 10.1161/CIRCEP.119.007811. Epub 2019 Nov 25. PMID 31760820
- [Result] Tu B, Wu L, Hu F, Fan S, Liu S, Liu L, Ding L, Zheng L, Yao Y. Cardiac deceleration capacity as an indicator for cardioneuroablation in patients with refractory vasovagal syncope. Heart Rhythm. 2022 Apr;19(4):562-569. doi: 10.1016/j.hrthm.2021.12.007. Epub 2021 Dec 9. PMID 34896621
- [Result] Zheng L, Sun W, Qiao Y, Hou B, Guo J, Killu A, Yao Y. Symptomatic Premature Ventricular Contractions in Vasovagal Syncope Patients: Autonomic Modulation and Catheter Ablation. Front Physiol. 2021 May 3;12:653225. doi: 10.3389/fphys.2021.653225. eCollection 2021. PMID 34012407
- [Result] Zheng L, Sun W, Liu S, Liang E, Du Z, Guo J, Wu L, Asirvatham SJ, Yao Y. The Diagnostic Value of Cardiac Deceleration Capacity in Vasovagal Syncope. Circ Arrhythm Electrophysiol. 2020 Dec;13(12):e008659. doi: 10.1161/CIRCEP.120.008659. Epub 2020 Nov 16. PMID 33197331
- [Result] Sun W, Zheng L, Qiao Y, Shi R, Hou B, Wu L, Guo J, Zhang S, Yao Y. Catheter Ablation as a Treatment for Vasovagal Syncope: Long-Term Outcome of Endocardial Autonomic Modification of the Left Atrium. J Am Heart Assoc. 2016 Jul 8;5(7):e003471. doi: 10.1161/JAHA.116.003471. PMID 27402231
- [Result] Wu L, Lu Y, Zheng L, Qiao YU, Chen G, Ding L, Hou B, Sun W, Liew R, Zhang S, Yao Y. Comparison of Radiofrequency Catheter Ablation Between Asymptomatic and Symptomatic Persistent Atrial Fibrillation: A Propensity Score Matched Analysis. J Cardiovasc Electrophysiol. 2016 May;27(5):531-5. doi: 10.1111/jce.12930. Epub 2016 Feb 12. PMID 26773415